CLINICAL TRIAL: NCT03111212
Title: Therapeutic Iloprost for the Treatment of Acute Respiratory Distress Syndrome (ARDS) (the ThIlo-Trial)
Brief Title: Iloprost in Acute Respiratory Distress Syndrome
Acronym: ThIlo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ThIlo
Record Dates: First submitted 2017-04-06; First posted 2017-04-12 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-06

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: Acute respiratory distress syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Iloprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Iloprost (Active Comparator)
  Interventions: Drug: Iloprost
- control (Placebo Comparator)
  Interventions: Drug: control

INTERVENTIONS:
Drug: Iloprost — Iloprost nebulized
  Arms: Iloprost
Drug: control — sodium chloride 0,9% nebulized
  Arms: control

SUMMARY:
The patients will be randomized into one of two groups. Both groups will receive standard care as is state of the art. The intervention group will receive Iloprost nebulized as inhalative therapy.

ELIGIBILITY:
Inclusion Criteria:

* Horowitz index <300
* Bilateral opacities on frontal chest radiograph
* requirement of positive pressure ventilation
* no clinical evidence of left atrial hypertension
* enrollment within 48h of onset of ARDS
* mechanical ventilation <7 days

Exclusion Criteria:

* age <18 years
* mechanical ventilation >7 days
* patient, surrogate or physician not committed to full intensive care support
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-08-14 (Actual)

PRIMARY OUTCOMES:
Oxygenation Index on Day 5 of Prostacyclin Treatment measured as PaO2/FiO2 | Day 6 of Study
  partial pressure of oxygen in blood (PaO2), in millimeters of mercury divided by the fraction of oxygen in the inhaled air (FiO2)

SECONDARY OUTCOMES:
Overall survival in 90-day follow-up period | on day 90 after randomization and study entry
  90 day all cause mortality
Sequential Organ Failure Assessment Score (SOFA Score) | until ICU discharge, estimated average = 14 days
  The SOFA score is based on six different scores, one each for the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems. Each system is assessed by 0=normal function to max 4 points=severe organ dysfunction Lowest Score is 0, the Maximums Score is 24; high Scores mean worse outcome
Duration of Mechanical Ventilation | until ICU discharge, estimated average = 14 days
  Ventilation Support length
Number of Patients with the Occurence of Barotrauma | until ICU discharge, estimated average = 14 days
  Barotrauma is damage to body tissue secondary to pressure difference in enclosed cavities within the body.Ventilator asynchrony, acute elevation of the plateau and peak pressures above 30 cmH2O, or sudden decrease of delivered tidal volume are result of barotrauma.
Number of Patients with Pulmonary Hemorrhage | until ICU discharge, estimated average = 14 days
  Significant Bleeding from Lung
Number of Patients with Gastrointestinal Hemorrhage | until ICU discharge, estimated average = 14 days
  Significant Bleeding from GI Tract
Number of Patients with Pulmonary Embolism | until ICU discharge, estimated average = 14 days
  Blockage of an artery in the lungs by a embolus that has moved from elsewhere in the body to the lung
Number of Patients with Delirium | until ICU discharge, estimated average = 14 days
  An organically caused decline from a previous baseline mental functioning, that develops over a short period of time, typically hours to days. Measured as occurence and length in time.
Number of Patients with ICU Acquired Weakness | until ICU discharge, estimated average = 14 days
  Skeletal muscle dysfunction
Discharge Location | until ICU discharge, estimated average = 14 days
  Number of Patients discharged to home without additional care (self-care), home with additional care (home health care) and other care facilities such as nursing homes. Measured as % of patients discharged to either of these locations.
Barthel Index (BI) | at 6 months after study inclusion
  Is a measure using an ordinal scale used to measure performance in activities of daily living (ADL). The original 10-item form of the BI consists of 10 common ADL activities including: feeding, bathing, grooming, dressing, bowel control, bladder control, toileting, chair transfer, ambulation and stair climbing. Items are rated in terms of whether individuals can perform activities independently, with some assistance, or are dependent (scored as 10, 5 or 0). Items are weighted according to the level of nursing care required.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rosenberger, MD, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University Hospital Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Haeberle HA, Calov S, Martus P, Serna-Higuita LM, Koeppen M, Goll A, Bernard A, Zarbock A, Meersch M, Weiss R, Mehrlander M, Marx G, Putensen C, Bakchoul T, Magunia H, Nieswandt B, Mirakaj V, Rosenberger P. Inhaled prostacyclin therapy in the acute respiratory distress syndrome: a randomized controlled multicenter trial. Respir Res. 2023 Feb 18;24(1):58. doi: 10.1186/s12931-023-02346-0. PMID 36805707
- [Derived] Haeberle H, Prohaska S, Martus P, Straub A, Zarbock A, Marx G, Zago M, Giera M, Koeppen M, Rosenberger P. Therapeutic iloprost for the treatment of acute respiratory distress syndrome (ARDS) (the ThIlo trial): a prospective, randomized, multicenter phase II study. Trials. 2020 Mar 4;21(1):242. doi: 10.1186/s13063-020-4163-0. PMID 32131881